CLINICAL TRIAL: NCT05528133
Title: Phase II Study of Genomically Guided Radiation Dose Personalization in the Management of Triple Negative Breast Cancer
Brief Title: Genomically Guided Radiation Therapy in the Management of Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21757
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: Breast Cancer; Genomically Guided Radiation
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Radiosensitivity Index optimized (Experimental): Participants will be assigned to optimized arm based on their RSI score. Participants will receive whole breast radiation therapy with or without regional lymph node irradiation as appropriate with or without a boost to the lumpectomy cavity.
  Interventions: Radiation: Genomically Guided Radiation Therapy
- Radiosensitivity Index not optimized (Active Comparator): Participants will receive standard of care whole breast radiation therapy with or without regional lymph node irradiation as appropriate with a boost to the lumpectomy cavity.
  Interventions: Radiation: Genomically Guided Radiation Therapy

INTERVENTIONS:
Radiation: Genomically Guided Radiation Therapy — Participants will receive treatment 5 days per week, in once daily fractions. The total dose will be 50 Gy in 25 fractions or 42.56 Gy in 16 fractions with or without a boost of 10 Gy in 5 fractions to the cavity.
  Arms: Radiosensitivity Index optimized
Radiation: Genomically Guided Radiation Therapy — Participants will receive treatment 5 days per week, in once daily fractions. The total dose will be 50 Gy in 25 fractions or 42.56 Gy in 16 fractions with a boost of 10 Gy in 5 fractions to the cavity.
  Arms: Radiosensitivity Index not optimized

SUMMARY:
The purpose of the study is to determine the feasibility of genomically guided radiation therapy (RT) in people with triple negative (HER2 negative, hormone receptor negative) breast cancer undergoing breast conservation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants should have undergone breast conservation therapy with a lumpectomy and axillary evaluation to consist of a sentinel node biopsy or axillary dissection
* Confirmation of Triple Negative (TN) breast cancer by tissue biopsy
* Adequate tissue to calculate RSI
* To fulfill the requirement of HER2- disease, a breast cancer must not demonstrate, at initial diagnosis or upon subsequent biopsy, overexpression of HER2 by either IHC or in-situ hybridization as defined by the ASCO / CAP Guidelines
* To fulfill the requirement of hormone receptor (HR)- disease, a breast cancer must express (<10%), by immunohistochemistry (IHC), the hormone receptors (estrogen receptor [ER] and progesterone receptor [PR]) as defined in the American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) Guidelines
* Life expectancy >16 weeks
* KPS ≥ 70
* Age ≥ 18 years
* Participants with surgery within 14 days should have recovered from all effects of the surgery and be cleared by their surgeon
* There is no limit on prior systemic therapies
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study
* Ability to sign an informed consent form, which can be signed by a family member or health care proxy. Informed consent must be given before study enrollment

Exclusion Criteria:

* Major surgery or significant traumatic injury that has not been recovered from 14 days before study initiation
* Women who are pregnant or breastfeeding
* Positive surgical margins
* History of allergy or hypersensitivity to any of the study drugs or study drug components
* Metastatic breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Local Control | At 3 Years
  Local control will be defined as lack of progression in the ipsilateral breast as documented by response assessment imaging

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 Years
  OS will be measured from the date of study initiation to the date of death due to any cause.
Progression Free Survival (PFS) | Up to 5 years
  PFS is measured from the date of first treatment to the date of first observation of PD or death due to any cause.
Distant Control | Up to 5 Years
  Distant control will be defined by lack of progression outside the irradiated treatment field
Quality of Life following Genomically Guided Dose Personalization | Up to 5 Years
  Quality of life (QOL) will be assessed through the completion of the Functional Assessment of Cancer Therapy for Breast Cancer questionnaire (FACT-B). This quality of life questionnaire contains questions from the FACT-General (G) questionnaire in the domains of physical, social/family, emotional, and functional well-being as well as additional questions pertaining to patients with breast cancer. The questionnaire will be completed at screening, during protocol therapy and at follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Morton Plant Hospital - Baycare Health System, Clearwater, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE